CLINICAL TRIAL: NCT02489253
Title: Incidence and Characteristics of Coronary Atherosclerosis in Asymptomatic Patients With Familial Hypercholesterolemia According to Monogenic Versus Polygenic Status
Brief Title: Atherosclerosis in Familial Hypercholesterolemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: RFH FH Study
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- polygenic hypercholesterolemia: patients with high cholesterol level where no mutation was found in their FH-causing genes and had to gene score in their six LDL-C raising gene score undergo a carotid ultrasound, a CT coronary angiogram and a blood test
  Interventions: Other: CT coronary angiogram and carotid ultrasound
- monogenic FH: patients with a mutation in FH-causing gene undergo a carotid ultrasound, a CT coronary angiogram and a blood test
  Interventions: Other: CT coronary angiogram and carotid ultrasound

INTERVENTIONS:
Other: CT coronary angiogram and carotid ultrasound — Scans in addition to routine clinical care

SUMMARY:
Familial hypercholesterolemia (FH) is a common inherited disorder with a frequency of 1 in 500 in the UK. Our aim is compare the carotid and coronary artery atherosclerosis in monogenic FH and polygenic hypercholesterolemia with means of a carotid ultrasound, a coronary CT angiogram and biochemical biomarkers.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a common inherited disorder with a frequency of 1 in 500 in the UK. Previous Studies showed that risk of heart attack in these patients is at least 50% higher in men and 30% higher in women compared to the general population as they have high blood cholesterol since birth. We propose to develop a screening model based on non-invasive visualisation of the heart blood vessels (coronary arteries) by CT scan, ultrasound of the neck vessels (carotid arteries) and blood tests to access the extend of cholesterol deposit in the blood vessels in these patients. Participants with confirmed diagnosis of FH would be recruited from FH database registry at Royal Free Hospital. They would have a CT coronary angiogram, an ultrasound of carotid arteries and a blood test. The study is divided into overlapping stages of recruitment and data collection and data analysis. If CT scan shows more than 70% obstruction in their coronary arteries, they would be offered a coronary angiogram and an intracoronary Optical Coherence Tomography for assessment of their blood vessel blockage.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must give written informed consent to participate in the study, Male and female subjects ≥ 18 years old, documentation of clinical diagnosis of familial Hypercholesterolemia

Exclusion Criteria:

* Estimated GFR <45, pregnant women, Atrial fibrillation or unstable heart rate, Established ischemic heart disease, previous Percutaneous Coronary Investigations (PCI) or Coronary Artery Bypass Surgery (CABG), Known allergy to iodine contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 monogenic FH and 50 polygenic hypercholesterolemia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
carotid Intima Media thickness measurement | 24 months
  done by carotid ultrasound to look for risk of atherosclerosis

CONTACTS AND LOCATIONS:
Overall Officials: Roby Rakhit, Study Director — University College Hospital and Royal Free Hospital
Locations (1):
- Royal Free Hospital, London, London, United Kingdom